CLINICAL TRIAL: NCT03138564
Title: An Effectiveness-Implementation Trial of SPIRIT in ESRD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Mi-Kyung Song, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00094859; 1R01NR017018-01 (NIH)
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: End Stage Renal Disease
Keywords: Nursing; Nephrology; Behavioral Research; Social Research
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — ligroin

STUDY DESIGN:
Intervention Model Description: Dialysis clinics are randomized to provide the intervention or usual care. Patients of those clinics will be given the opportunity to participate in the study and will receive the intervention or usual care based on which clinic they attend.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPIRIT Clinic (Experimental): Patients at clinics that have been randomized to the SPIRIT arm will be given the option to participate in the intervention. SPIRIT is a two-session, 60-minute, structured psychoeducational intervention, targeting both patient and surrogate. Using a provider manual, the care provider follows six steps: 1) assessing illness presentation, 2) identifying gaps and concerns, 3) creating conditions for conceptual change, 4) introducing replacement information, 5) summarizing, and 6) setting goals and planning.
  Interventions: Behavioral: SPIRIT
- Comparison Condition Clinic (Active Comparator): Patients at clinics that have been randomized to the control arm will be given the option to participate as a study control. The control clinics will have delayed implementation of the SPIRIT intervention.
  Interventions: Behavioral: Comparison Condition

INTERVENTIONS:
Behavioral: SPIRIT — SPIRIT is a two-session, structured psychoeducational intervention assisting patients clarify their end-of-life preferences and helping surrogates understand the patient's wishes and prepare for the surrogate role.
  During the first session (about 45 minutes) individualized information is provided about the effectiveness of life-sustaining treatment for people with end-organ failure, and the care provider will assist the patient to examine his/her values about life-sustaining treatment. The surrogate will receive help preparing for end-of-life decision-making and the emotional burden of decision-making. A Goals-of-Care document will be completed to indicate the patient's preferences.
  Two weeks later, the second session (about 15 minutes) addresses remaining or new concerns. The patient's Goals-of-Care document will be reviewed. The patient's end-of-life preferences and surrogate's name and relationship to the patient will be documented in the medical record.
  Other Names: Sharing Patient's Illness Representation to Increase Trust
  Arms: SPIRIT Clinic
Behavioral: Comparison Condition — As required by Centers for Medicare and Medicaid Services (CMS), written information on advance directives (ADs) is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an AD. This typically takes about 10 minutes.
  Other Names: Usual care
  Arms: Comparison Condition Clinic

SUMMARY:
Despite advances in dialysis, only 50% of dialysis patients are alive 3 years after the onset of end-stage renal disease (ESRD). Although withdrawal of dialysis precedes 1 in 4 deaths of patients with ESRD, withdrawal from dialysis and aggressive treatment is rarely discussed by patients and their surrogates with sufficient time to consider alternatives such as hospice or dying at home. Over the last decade, the researchers have developed and iteratively tested a patient and family-centered advance care planning intervention based on the Representational Approach to Patient Education called "Sharing Patient's Illness Representation to Increase Trust" (SPIRIT). SPIRIT is a 6-step, 2-session, face-to-face intervention to promote cognitive and emotional preparation for end-of-life decision making for patients with ESRD and their surrogates.

This study is a multicenter, clinic-level cluster randomized trial to evaluate the effectiveness of SPIRIT delivered by dialysis care providers as part of routine care in free-standing outpatient dialysis clinics compared to usual care plus delayed SPIRIT implementation. The researchers will recruit 400 dyads of patients at high risk of death in the next year and their surrogates from dialysis clinics in four states. Patients and surrogates will complete questionnaires at baseline and two weeks after the intervention. Surrogates will complete a post-bereavement assessment three months after the death of the patient.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) currently affects nearly 662,000 people in the U.S. While dialysis is the treatment of choice for over 90% of patients with ESRD and is universally covered by Medicare regardless of patient age or means, the likelihood that dialysis can restore health or prolong life is limited; only 50% of dialysis patients are alive 3 years after the onset of ESRD. Thus many dialysis patients and their family members or surrogate decision-makers have to face difficult end-of-life decisions. Although advance care planning (ACP), in which patients and surrogate decision-makers discuss future health states and treatment options, is a central tenet of dialysis care, the vast majority of dialysis patients (>90%) report never engaging in ACP discussions with their care providers. The lack of effective ACP to prepare patients and their surrogates for end-of-life decision making with sufficient time before death has deleterious consequences at all levels of society. Consequences have been well documented: prolonged use of futile treatment at the end of life, which misuses the healthcare system, high levels of surrogate distress during decision making, which emanates from not having a clear understanding of the patient's wishes, and surrogates experiencing later sequelae of psychosocial morbidities, such as depression and family discord.

"Sharing Patient's Illness Representation to Increase Trust" (SPIRIT), a patient and family-centered ACP intervention based on the Representational Approach to Patient Education, was designed by the research team to establish a testable model of how end-of-life care discussions could occur between a dialysis patient and his/her chosen surrogate (usually a spouse or adult child). The discussions, which are facilitated by a trained care provider, are framed around addressing each individual's representations of (beliefs about) the illness and views of life-sustaining measures at the end of life. SPIRIT follows a six-step learning objective over two-sessions, which together take about 60 minutes. The care provider, who is value-neutral, guides the patient in examining his/her values related to end-of-life care, helps the surrogate understand the patient's illness progression, and prepares the surrogate for his/her role as a surrogate in a highly emotionally charged medical setting. Over the last decade, SPIRIT has been tested to establish feasibility, patient-surrogate acceptability, and efficacy. In these explanatory trials carried out in dialysis clinics, SPIRIT was delivered by trained research nurses. Patients and surrogates in SPIRIT showed significant improvement in preparedness for end-of-life decision making, including the extent to which: a) the patient and surrogate agreed on end-of-life care goals, b) the patient had reduced conflict about the benefits and burdens of life-sustaining treatments, and c) the surrogate had increased confidence about the role of surrogate. Key to establishing the utility of this approach for broader generalizability, surrogates who received SPIRIT reported significantly improved post-bereavement psychological outcomes after the patient's death compared to those who did not. The logical, critical next step is to ask: Will SPIRIT be effective as part of routine care in real-world clinical settings with less control? To address this very issue, the researchers will conduct a real-world effectiveness-implementation study, an essential step prior to widespread implementation of SPIRIT.

This study is a multicenter, clinic-level cluster randomized trial to evaluate the effectiveness of SPIRIT delivered by dialysis care providers as part of routine care in free-standing outpatient dialysis clinics compared to usual care plus delayed SPIRIT implementation. Simultaneously, the researchers will evaluate the implementation of SPIRIT, including sustainability. This study will use a Type I effectiveness-implementation hybrid approach that combines testing intervention effectiveness and gathering information about implementation of an efficacious intervention in a real world setting. To maximize data on the implementation process and sustainability, the researchers chose a delayed intervention design in which clinics are randomized either to implement SPIRIT immediately after randomization (i.e., initial implementation) or to maintain usual care for a comparison condition and then implement the intervention in control clinics following conclusion of this clinical trial (i.e., delayed implementation). The intent of the delayed implementation group was provide descriptive data for translation of the intervention into clinical practice (versus data collected on dyad participants in this current study), however, this portion of the study could not be performed due to the coronavirus disease 2019 (COVID-19) pandemic.

The short-term goal is to generate sufficient evidence to accelerate the integration of SPIRIT into dialysis practice and policy. This study will recruit 400 dyads of patients at high risk of death in the next year and their surrogates (a total of 800 individuals) from dialysis clinics in four states. The dialysis clinics will be randomized to implement SPIRIT or to maintain usual care to serve as a control to the intervention. Participants will complete a follow-up assessment two weeks after the the study intervention. They will then be observed for 9 months (or until the death of the patient) with an optional extension of the observational period for an additional 12 months, for up to 21 months of observation. Individual patient participation will end after the observation period (9 or 21 months) or death, whichever occurs first; surrogate participation will end after the observation period (9 or 21 months) or at the completion of the post-bereavement surveys which are administered 3-months after the death of the patient (up to 24 months).

ELIGIBILITY:
Inclusion Criteria for Patients:

* on either hemodialysis or peritoneal dialysis
* able to understand and speak English

Exclusion Criteria for Patients:

* lack of an available surrogate
* too ill or cognitively impaired to participate based on clinicians' judgment
* already enrolled in hospice

Inclusion Criteria for Surrogates:

* are chosen as a surrogate by the patient
* paid caregivers who will not be participating in medical decisions for the patient

Exclusion Criteria for Surrogates:

* Unable to complete questionnaires due to physical or cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mi-Kyung Song, PhD, RN, Principal Investigator — Emory University
Locations (39):
- United States (39):
  - Emory Dialysis at Northside, Atlanta, Georgia
  - Emory Dialysis at Greenbriar, Atlanta, Georgia
  - Emory Dialysis at Candler, Decatur, Georgia
  - Emory Dialysis Center, North Decatur, Georgia
  - Dialysis Clinic, Inc - Acoma Canoncito Laguna, Acoma Pueblo, New Mexico
  - Dialysis Clinic, Inc - Albuquerque, Albuquerque, New Mexico
  - Dialysis Clinic, Inc - Albuquerque South, Albuquerque, New Mexico
  - Dialysis Clinic, Inc - Albuquerque East, Albuquerque, New Mexico
  - Dialysis Clinic, Inc - Carlsbad, Carlsbad, New Mexico
  - Dialysis Clinic, Inc - Cuba, Cuba, New Mexico
  - Dialysis Clinic, Inc - Grants, Grants, New Mexico
  - Dialysis Clinic, Inc - Raton, Raton, New Mexico
  - Dialysis Clinic, Inc - Rio Rancho, Rio Rancho, New Mexico
  - Dialysis Clinic, Inc - Santo Domingo, Santo Domingo Pueblo, New Mexico
  - Dialysis Clinic, Inc - Silver City, Silver City, New Mexico
  - Dialysis Clinic, Inc - Taos, Taos, New Mexico
  - Carolina Dialysis - Carrboro, Carrboro, North Carolina
  - Carolina Dialysis - Mebane, Mebane, North Carolina
  - Carolina Dialysis - Pittsboro, Pittsboro, North Carolina
  - Fresenius Kidney Care - Raleigh, Raleigh, North Carolina
  - Carolina Dialysis-Sanford Lee County, Sanford, North Carolina
  - Carolina Dialysis-Sanford Main, Sanford, North Carolina
  - Carolina Dialysis - Siler City, Siler City, North Carolina
  - Dialysis Clinic, Inc - Harmar Village, Cheswick, Pennsylvania
  - Dialysis Clinic, Inc - Monroeville/Five Points, Monroeville, Pennsylvania
  - Dialysis Clinic, Inc - North Versailles, North Versailles, Pennsylvania
  - Dialysis Clinic, Inc - Oakland, Pittsburgh, Pennsylvania
  - Dialysis Clinic, Inc - Banksville, Pittsburgh, Pennsylvania
  - Dialysis Clinic, Inc - Wilkinsburg, Pittsburgh, Pennsylvania
  - Dialysis Clinic, Inc - North Hills, Pittsburgh, Pennsylvania
  - UVA Dialysis Altavista Clinic, Altavista, Virginia
  - UVA Dialysis Amherst Clinic, Amherst, Virginia
  - Kidney Center Outpatient Dialysis Clinic, Charlottesville, Virginia
  - UVA Dialysis Clinic Farmville, Farmville, Virginia
  - UVA Augusta Dialysis, Fishersville, Virginia
  - UVA Dialysis Zion Crossroads, Gordonsville, Virginia
  - UVA Dialysis Lynchburg, Lynchburg, Virginia
  - UVA Dialysis Orange Clinic, Orange, Virginia
  - UVA Dialysis Clinic Staunton, Staunton, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song MK, Unruh ML, Manatunga A, Plantinga LC, Lea J, Jhamb M, Kshirsagar AV, Ward SE. SPIRIT trial: A phase III pragmatic trial of an advance care planning intervention in ESRD. Contemp Clin Trials. 2018 Jan;64:188-194. doi: 10.1016/j.cct.2017.10.005. Epub 2017 Oct 6. PMID 28993286
- [Derived] Song MK, Manatunga A, Plantinga L, Metzger M, Kshirsagar AV, Lea J, Abdel-Rahman EM, Jhamb M, Wu E, Englert J, Ward SE. Effectiveness of an Advance Care Planning Intervention in Adults Receiving Dialysis and Their Families: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2351511. doi: 10.1001/jamanetworkopen.2023.51511. PMID 38289604

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from multiple dialysis centers in Georgia, New Mexico, North Carolina, Pennsylvania, and Virginia, USA. Participant enrollment began on February 15, 2018, and follow-up assessments for the primary outcome measures at Week 2 were completed on March 24, 2022. Data collection for secondary outcome measures with surrogates three months after the patient's death was completed July 29, 2022.
Pre-assignment Details: 42 clinics were enrolled with 23 randomized to the SPIRIT and 19 randomized to usual care. One SPIRIT clinic and 2 control clinics were excluded prior to study initiation. There were 557 eligible patients in SPIRIT clinics and 264 dyads consented to participate; of these, 33 dyads withdrew or became ineligible prior to the baseline visit. In control clinics there were 293 eligible patients and 210 dyads consented to participate; 15 dyads withdrew or became ineligible prior to the baseline visit.
Units Other Than Participants: dialysis clinics
Groups:
- SPIRIT Clinic: Dialysis clinics randomized to deliver the SPIRIT intervention. SPIRIT is a two-session, 60-minute, structured psychoeducational intervention, targeting both patient and surrogate. Using a provider manual, the care provider follows six steps: 1) assessing illness presentation, 2) identifying gaps and concerns, 3) creating conditions for conceptual change, 4) introducing replacement information, 5) summarizing, and 6) setting goals and planning.
  Patients receiving care at SPIRIT clinics were given the option to participate in this study with their surrogate decision-makers.
- Comparison Condition Clinic: Dialysis clinics randomized to the comparison condition control arm.
  The comparison condition is the usual care provided. As required by the Centers for Medicare and Medicaid Services (CMS), written information on advance directives (ADs) is provided to a patient on the first day of dialysis, and a social worker reviews this information with patients and encourages them to complete an AD. This typically takes about 10 minutes.
  Patients receiving care at the comparison condition clinics were given the option to participate in this study with their surrogate decision-makers.
Period: Overall Study
Arm/Group | SPIRIT Clinic | Comparison Condition Clinic
Started | 462; 22 dialysis clinics | 390; 17 dialysis clinics
Patients Beginning the Study | 231; 22 dialysis clinics | 195; 17 dialysis clinics
Surrogates Beginning the Study | 231; 22 dialysis clinics | 195; 17 dialysis clinics
Patients Completing the Week 2 Assessment | 182; 22 dialysis clinics | 192; 17 dialysis clinics
Surrogates Completing the Week 2 Assessment | 183; 22 dialysis clinics | 189; 17 dialysis clinics
Surrogates Eligible for Post-bereavement Visit | 54; 22 dialysis clinics | 35; 17 dialysis clinics
Surrogates Completing Post-bereavement Visit | 46; 22 dialysis clinics | 31; 17 dialysis clinics
Completed (Completed Week 2 visit) | 365; 22 dialysis clinics | 381; 17 dialysis clinics
Not Completed | 97; 0 dialysis clinics | 9; 0 dialysis clinics
Not completed — Death of patient prior to the Week 2 assessment | 14 | 2
Not completed — Lost to Follow-up | 16 | 2
Not completed — Withdrawal by Subject | 48 | 4
Not completed — No longer met eligibility criteria | 2 | 0
Not completed — Withdrawal by investigator due to no availability of SPIRIT champion in the clinic | 4 | 0
Not completed — Patient died before surrogate completed Week 2 assessment | 12 | 0
Not completed — Surrogate declined to complete the Week 2 assessment but did not withdraw from study | 0 | 1
Not completed — Death of surrogate prior to Week 2 assessment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- SPIRIT Clinic - Patients: Patients receiving care at clinics randomized to the SPIRIT intervention
- SPIRIT Clinic - Surrogates: Surrogates of patients receiving care at clinics randomized to the SPIRIT intervention
- Comparison Condition Clinic - Patients: Patients receiving care at clinics randomized to the control condition
- Comparison Condition Clinic - Surrogates: Surrogates of patients receiving care at clinics randomized to the control condition
- Total: Total of all reporting groups
Arm/Group | SPIRIT Clinic - Patients | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Patients | Comparison Condition Clinic - Surrogates | Total
Number analyzed (Participants) | 231 | 231 | 195 | 195 | 852
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (12.8) | 53.2 (14.7) | 62.4 (12.5) | 54.3 (16.1) | 57.8 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 168 | 97 | 152 | 538
  Male | 110 | 63 | 98 | 43 | 314
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 5 | 8 | 28
  Not Hispanic or Latino | 222 | 225 | 190 | 185 | 822
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 3 | 1 | 6
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 161 | 159 | 132 | 132 | 584
  White | 66 | 64 | 53 | 57 | 240
  More than one race | 2 | 4 | 4 | 1 | 11
  Unknown or Not Reported | 0 | 2 | 3 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 231 | 231 | 195 | 195 | 852

OUTCOME MEASURES:

1. Primary Outcome: Dyad Congruence on Goals-of-Care Tool
Description: The Goals-of-Care Tool which includes two scenarios describing medical conditions commonly occurring in end-stage renal disease (ESRD) patients. Possible responses to the scenarios are: "The goals of care should focus on delaying my death, and thus I want to continue life-sustaining treatment", "The goals of care should focus on my comfort and peace, and thus I do not want life-sustaining treatment, including dialysis", and "I am not sure". Patients and surrogates complete this tool independently and their responses are compared to determine dyad congruence. A dyad is assigned with "1" if each member of the dyad chose the same response (either comfort care only or continue aggressive care) in both scenarios. In all other cases, the dyad is assigned with "0", which includes: 1) the patient and surrogate responses are the same in one of the two scenarios, 2) the patient and surrogate responses differ in both scenarios, and 3) the patient and surrogate responses are both "I am not sure".
Time Frame: Baseline, Week 2
Population: The number of participants analyzed reflects the number of persons with ESRD and surrogate dyads (two persons per dyad). This analysis includes dyads who both completed the assessment at the indicated study visit.
Measure: Number; unit: dyads
Groups:
- SPIRIT Clinic - Dyads: Patient and surrogate dyads at clinics randomized to the SPIRIT intervention
- Comparison Condition Clinic - Dyads: Patient and surrogate dyads at clinics randomized to the control condition
Arm/Group | SPIRIT Clinic - Dyads | Comparison Condition Clinic - Dyads
Number analyzed (Participants) | 231 | 195
dyads
  Number of Congruent Dyads at Baseline (assigned value = 1) | 98 | 76
  Number of Incongruent Dyads at Baseline (assigned value = 0) | 133 | 119
  Number of Congruent Dyads at 2 Weeks Post-Intervention (assigned value = 1): number analyzed (Participants) | 182 | 187
  Number of Congruent Dyads at 2 Weeks Post-Intervention (assigned value = 1) | 111 | 94
  Number of Incongruent Dyads at 2 Weeks Post-Intervention (assigned value = 0): number analyzed (Participants) | 182 | 187
  Number of Incongruent Dyads at 2 Weeks Post-Intervention (assigned value = 0) | 71 | 93

2. Primary Outcome: Patient's Decisional Conflict Scale (DCS) Score
Description: Patient decisional conflict is measured using the 13-item Decisional Conflict Scale (DCS), a validated measure in the context of end-of-life decision making. Participants indicate their level of agreement with statements about their plans for their future medical care by selecting (1) Strongly Agree, (2) Agree, (3) Neither Agree nor Disagree, (4) Disagree, or (5) Strongly Disagree. The total score ranges from 13 to 65 with higher scores indicating greater difficulty in weighing benefits and burdens of life-sustaining treatments and decision making.
Time Frame: Baseline, Week 2
Population: This analysis includes patient participants who completed the DCS. One participant in the comparison condition study arm did not answer all items on the scale at the baseline visit and thus their total score could not be computed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Clinic - Patients | Comparison Condition Clinic - Patients
Number analyzed (Participants) | 231 | 194
score on a scale
  Baseline | 25.6 (6.22) | 24.8 (5.82)
  Two Weeks Post-Intervention: number analyzed (Participants) | 182 | 192
  Two Weeks Post-Intervention | 23.4 (5.94) | 24.1 (5.78)

3. Primary Outcome: Surrogate's Decision Making Confidence (DMC) Scale Score
Description: Surrogate decision-making confidence is measured using the 5-item Decision Making Confidence (DMC) scale. Surrogates indicate how confident they are about making medical decisions if the patient becomes unable to make their own decisions by their level of agreement with statements along a scale of (0) "Not confident at all" to (4) "Very confident". Total scores range from 0 to 20, with higher scores indicating greater confidence.
Time Frame: Baseline, Week 2
Population: This analysis includes participants completing the indicated study visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Surrogates
Number analyzed (Participants) | 231 | 195
Score on a scale
  Baseline | 18.2 (2.73) | 18.3 (2.59)
  Two Weeks Post-Intervention: number analyzed (Participants) | 183 | 189
  Two Weeks Post-Intervention | 18.9 (1.73) | 18.6 (2.16)

4. Primary Outcome: Composite Outcome of Dyad Congruence and Surrogate DMC Score
Description: The composite outcome combines dyad congruence on Goals-of-Care scenarios and surrogate DMC scores. If the dyad congruence is 1 and the surrogate's DMC >=3, then the composite outcome value for the dyad is "1". In all other cases, the dyad's composite outcome value is "0".
Time Frame: Baseline, Week 2
Population: The number of participants analyzed reflects the number of persons with ESRD and surrogate dyads (two persons per dyad). This analysis includes dyads who both completed the assessments at the indicated study visit.
Measure: Number; unit: dyads
Arm/Group | SPIRIT Clinic - Dyads | Comparison Condition Clinic - Dyads
Number analyzed (Participants) | 231 | 195
dyads
  Number of Dyads Where Baseline Composite Outcome = 1 | 92 | 74
  Number of Dyads Where Baseline Composite Outcome = 0 | 139 | 121
  Number of Dyads Where Week 2 Post-Intervention Composite Outcome = 1: number analyzed (Participants) | 182 | 187
  Number of Dyads Where Week 2 Post-Intervention Composite Outcome = 1 | 107 | 90
  Number of Dyads Where Week 2 Post-Intervention Composite Outcome = 0: number analyzed (Participants) | 182 | 187
  Number of Dyads Where Week 2 Post-Intervention Composite Outcome = 0 | 75 | 97

5. Secondary Outcome: End-of-life Treatment Intensity
Description: The use of intensive procedures during end-of-life treatment will be identified through the United States Renal Data System (USRDS). The use of mechanical ventilation as part of the patient's end-of-life (EOL) treatment will be documented (e.g., mechanical ventilation, feeding tube, dialysis, CPR). The EoL treatment intensity data acquisition will take at least two more years after the participant's death due to the 2-year gap in the administrative data release.
Time Frame: Upon patient death (up to 21 months)
Reporting Status: Not Posted, anticipated posting 2026-03

6. Secondary Outcome: Surrogate's Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: Surrogate post-bereavement anxiety symptoms were measured with the Hospital Anxiety and Depression Scale (HADS) Anxiety subscale. Surrogates indicate their level of agreement with statements by selecting responses rated from 0 (the problem in the statement is not an issue) to 3 (the problem in the statement is a very big issue). Scores for the anxiety subscale range from 0 to 21 with higher scores indicating greater symptom severity. A score of 0-7 indicates "normal", 8-10 indicates "borderline abnormal", and 11-21 indicates "abnormal" levels of anxiety.
Time Frame: Baseline, 3 months after patient death (up to 24 months)
Population: This analysis includes surrogates from dyads where the patient died during the follow-up period. Per the intent to treat analysis, surrogates of 89 deceased patients were to be analyzed, and baseline values are presented for these participants. Twelve did not complete the post-bereavement survey due to being lost to follow-up or not consenting to participate in the extended follow-up. Baseline and post-bereavement scores are presented for the 77 who completed the post-bereavement assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Surrogates
Number analyzed (Participants) | 54 | 35
score on a scale
  Baseline for all surrogates where the patient died during the follow-up period | 4.80 (2.99) | 4.89 (2.83)
  Baseline for surrogates who completed the post-bereavement assessment: number analyzed (Participants) | 46 | 31
  Baseline for surrogates who completed the post-bereavement assessment | 4.85 (3.07) | 4.61 (2.81)
  Post-bereavement assessment (3 months after patient death): number analyzed (Participants) | 46 | 31
  Post-bereavement assessment (3 months after patient death) | 5.59 (3.58) | 6.71 (3.72)

7. Secondary Outcome: Surrogate's Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: Surrogate post-bereavement symptoms of depression were measured with the Hospital Anxiety and Depression Scale (HADS) Depression subscale. Surrogates indicate their level of agreement with statements by selecting responses rated from 0 (the problem in the statement is not an issue) to 3 (the problem in the statement is a very big issue). Total scores of the depression subscale range from 0 to 21 with higher scores indicating greater symptom severity. A score of 0-7 indicates "normal", 8-10 indicates "borderline abnormal", and 11-21 indicates "abnormal" levels of depression.
Time Frame: Baseline, 3 months after patient death (up to 24 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Surrogates
Number analyzed (Participants) | 54 | 35
score on a scale
  Baseline for all surrogates where the patient died during the follow-up period | 3.28 (2.62) | 2.83 (2.80)
  Baseline for surrogates who completed the post-bereavement assessment: number analyzed (Participants) | 46 | 31
  Baseline for surrogates who completed the post-bereavement assessment | 3.04 (2.36) | 2.71 (2.76)
  Post-bereavement assessment (3 months after patient death): number analyzed (Participants) | 46 | 31
  Post-bereavement assessment (3 months after patient death) | 4.26 (2.94) | 4.23 (2.69)

8. Secondary Outcome: Surrogate's Post-Traumatic Symptoms Scale-10 (PTSS-10) Score
Description: Surrogate post-bereavement traumatic distress was measured with the Post-Traumatic Symptoms Scale-10 (PTSS-10). Surrogates indicate how often they have experienced symptoms of post-traumatic stress by responding to 10 symptoms on a scale of 1 to 7 where 1 = "never" and 7 = "always". Total scale scores range from 10 to 70 and higher scores indicate more intense symptoms.
Time Frame: Baseline, 3 months after patient death (up to 24 months)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Surrogates
Number analyzed (Participants) | 54 | 35
score on a scale
  Baseline for all surrogates where the patient died during the follow-up period | 19.96 (9.24) | 21.97 (9.87)
  Baseline for surrogates who completed the post-bereavement assessment: number analyzed (Participants) | 46 | 31
  Baseline for surrogates who completed the post-bereavement assessment | 19.30 (7.81) | 21.97 (10.26)
  Post-bereavement assessment (3 months after patient death): number analyzed (Participants) | 46 | 31
  Post-bereavement assessment (3 months after patient death) | 26.4 (12.2) | 29.3 (13.3)

ADVERSE EVENTS:
Time Frame: Adverse events were documented during the intervention session (Day 1). Dyads remained in the study to be followed for patient deaths for 9 months and after that they could opt to be followed for an additional 12 months, for up to 21 months in total. When a patient died the surrogate was asked to complete a post-bereavement assessment 3 months after the patient death, and then their study participation was considered complete (up to 24 months).
Description: Only adverse events related to the intervention, such as emotional distress, were documented during the intervention session. Patient deaths are reported in the mortality table, however, due to the population being examined and the nature of this study, deaths among patients with ESRD are not considered to be adverse events of the study. Patient deaths were collected to assess post-bereavement outcomes among surrogates.
Arm/Group | SPIRIT Clinic - Patients | SPIRIT Clinic - Surrogates | Comparison Condition Clinic - Patients | Comparison Condition Clinic - Surrogates
All-Cause Mortality (participants affected / at risk) | 54/231 | 1/231 | 35/195 | 0/195
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/231 | 0/195 | 0/195
Other Adverse Events (participants affected / at risk) | 0/231 | 0/231 | 0/195 | 0/195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT03138564/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT03138564/ICF_001.pdf